CLINICAL TRIAL: NCT04000126
Title: Pupillometry - Future of Objective Pain Reaction Measurement While Unconscious
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury (Other)
Responsible Party: Principal Investigator, Malgorzata Braczkowska, Principal Investigator, University of Warmia and Mazury
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UWarmiaMazury
Record Dates: First submitted 2019-05-01; First posted 2019-06-27 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pain
Keywords: lidocaine; intubation; pupillometry; hemodynamic response; pain; reflex; pupillary monitoring; intraoperative; analgesia; general anesthesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine; Sodium Chloride; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control C (Active Comparator): This group will be given induction anesthesia agents in standard doses (fentanyl 3mcg/kg, propofol 2mg/ kg, rocuronium 0,6mg/kg)
  Interventions: Device: Pupil reflex dilation measurement (PRD); Device: PPI (Pupillary Pain Index); Device: Bispectral Index (BIS); Device: HR; Device: BP
- Lignocaine group L (Experimental): This group will be given additionally 1.5 mg/kg lidocaine/ 100ml 0,9% NaCl iv 10min before intubation
  Interventions: Device: Pupil reflex dilation measurement (PRD); Device: PPI (Pupillary Pain Index); Drug: lidocaine; Device: Bispectral Index (BIS); Device: HR; Device: BP
- Placebo P (Placebo Comparator): This group will be given additionally 100 ml 0,9% NaCl iv 10 min before intubation
  Interventions: Device: Pupil reflex dilation measurement (PRD); Device: PPI (Pupillary Pain Index); Drug: Placebo; Device: Bispectral Index (BIS); Device: HR; Device: BP

INTERVENTIONS:
Device: Pupil reflex dilation measurement (PRD) — Pupillary Reflex Dilation (PRD) measured for 60 s during orotracheal intubation using a video pupillometer
Device: PPI (Pupillary Pain Index) — Pupillary Reflex Dilation (PRD) measured using a video pupillometer 5 min after orotracheal intubation
Drug: lidocaine — 1.5 mg/kg lidocaine/ 100ml 0,9% NaCl iv 10min before intubation
  Other Names: lidocaine, Xylocaine
  Arms: Lignocaine group L
Drug: Placebo — 100ml 0,9% NaCl iv 10min before intubation
  Other Names: 0,9% natrium chloratum, sodium chloride
  Arms: Placebo P
Device: Bispectral Index (BIS) — Bispectral Index will be monitored to assess the depth of anaesthesia
Device: HR — HR in beats/min will be measured by the electrocardiogram monitor
Device: BP — BP will be measured automatically by an occluding upper arm cuff

SUMMARY:
This study aims to assess the usefulness of pupillometry as a nociceptive indicator during elective orotracheal intubation in patients given intravenous lignocaine pre-intubation as compared to a placebo pre-intubation.

DETAILED DESCRIPTION:
Laryngoscopy and tracheal intubation are associated with a sympathetic discharge caused by stimulation of the upper respiratory tract. Venous lidocaine is the agent most used to attenuate the hemodynamic response to laryngoscopy and intubation. Hemodynamic response might be masked by the drugs the patient is taking and its status (ex. sepsis). There's a need for an objective pain assessment method while the patient is unconscious, to maintain a proper level of analgesia and to control the hemodynamic response in order to decrease systemic repercussions.

This single-blind, randomized, single center, prospective study was approved by the Bioethics Committee of the University of Warmia and Mazury under the report number 11/2019 21st of February 2019.

Patients scheduled for elective surgery under general anesthesia with tracheal intubation were divided into three groups:

Group 1: anaesthetic induction with standard doses iv was performed (fentanyl 3mcg/kg, propofol 2mg/kg, rocuronium 0,6mg/kg).

Group 2: same as in group 1 + lidocaine 1,5mg/kg w 100ml 0,9% NaCl 10 min before intubation.

Group 3 (placebo group): same as group 1 + 100ml 0,9% NaCl 10 min before intubation

The values for blood pressure (NIBP), heart rate (HR), Train of four (TOF) and bispectral index (BIS) were measured in all groups during the whole time of the protocol. PRD (Pupillary Reflex Dilation) was measured in the exact time of intubation. Additionally, after intubation PPI (Pupillary Pain Index) was checked.

During the whole protocol BIS value was maintained to be equal to or less than 50, if this value was not reached, a venous increment of 1mg/kg of propofol was administered.

Hypertension was considered when the BP values were 20% above baseline values or if Systolic Blood Pressure (SBP) > 140 mmHg. Hypotension was considered when the Blood Pressure (BP) values were 20% below baseline values or if SBP > 90 mmHg. Tachycardia was considered when the Heart Rate (HR) values were 20% above baseline values or if HR > 100 mmHg. Bradycardia was considered for HR values under 50 bpm.

ELIGIBILITY:
Inclusion Criteria:

* Physical State 1 or 2 of the American Society of Anesthesiology (ASA)
* Electively scheduled for surgery requiring general anesthesia
* Age >18 years

Exclusion Criteria:

* Difficult airway
* Unanticipated difficult airway based on the previous history of difficult intubation
* Urgently scheduled for surgery requiring general anesthesia
* Ophthalmologic pathology precluding pupillometry, ex. Horner's syndrome, Sjogrens syndrome
* Anisocoria
* History of opioid abuse
* Subjects who are or may be pregnant
* Unable to converse in Polish
* History of psychiatric/cognitive disease
* Patients who do not give informed consent
* Patients with contraindications or history of hypersensitivity to lidocaine
* Patients with coronary ischemic disease
* Patients with atrioventricular block at any grade
* Patients with diagnosed cardiac arrhythmias
* Patients with heart failure
* Patients who are taking drugs influencing the pupil size
* Patients with pacemaker
* Patients younger than 18 years of age
* History of chronic pain, chronic opioid use (> 3 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Usefulness of Pupillary Reflex Dilation (PRD) measured using a video pupillometer in determining the role of lidocaine iv before intubation. | PRD: during the exact time of intubation (continuous measurement for 60 seconds)
  Level of analgesia will be investigated in all groups (placebo, lidocaine, control) basing on the autonomous system activation during intubation by measuring variation of pupil diameter (% and mm).

SECONDARY OUTCOMES:
The influence of intravenous lidocaine on level of analgesia during orotracheal intubation | PRD: during the exact time of intubation (continuous measurement for 60 seconds)
  Changes that occur in PRD measured using video pupillometer as a response to an analgesic intervention will be investigated in all groups (placebo, lidocaine, control).
The influence of intravenous lidocaine on level of analgesia during orotracheal intubation. | HR - baseline and 0,1,2,3,4 minutes post-intubation
  Level of analgesia will be investigated in all groups (placebo, lidocaine, control) basing on the autonomous system activation during intubation by measuring changes in HR (beats/min)
The influence of intravenous lidocaine on level of analgesia during orotracheal intubation. | BP - baseline and 0,1,2,3,4 minutes post-intubation
  Level of analgesia will be investigated in all groups (placebo, lidocaine, control) basing on the autonomous system activation during intubation by measuring changes in BP (mmHg)
Correlation between PRD and PPI (Pupillary Pain Index) measured using video pupillometer and BIS (Bispectral Index) | BIS - baseline, during intubation, 0,1,2,3,4,5 minutes post-intubation, PRD: during the exact time of intubation (continuous measurement for 60 seconds), PPI - 5 minutes post-intubation
  Changes that occur in PRD and PPI as a response to an analgesic intervention will be investigated in all groups (placebo, lidocaine, control) and correlated to BIS in all groups.
The influence of intravenous lidocaine on PPI | 5 minutes post-intubation
  Changes that occur in PPI measure using video pupillometer as a response to an analgesic intervention will be investigated in all groups (placebo, lidocaine, control).

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Mayzner-Zawadzka, MD,PhD,Prof, Study Chair — Anesthesiology and Intensive Care Clinical Ward, University of Warmia and Mazury
Locations (1):
- Anesthesiology and Intensive Care Clinical Ward, Clinical University Hospital, Olsztyn, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified study participants data for all primary and secondary outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data will be made available for researchers who provide a methodologically sound proposal. Proposals should be directed to m.braczkowska@gmail.com . Data access requests will be reviewed by an External Independent Review Panel. To gain access, data requestors will need to sign a data access agreement.